CLINICAL TRIAL: NCT02893449
Title: Improvement of Social Adaptation After Pre-operative Cognitive Remediation in Parkinson's Patients Profiting From a Bilateral Subthalamic Stimulation
Brief Title: Psychiatry Study: Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PSY PARKINSON
Record Dates: First submitted 2010-02-05; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson; SAS-SR; Social adaptation; Patients suffering from Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Social Adjustment | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SICRPPD group (Other): (Specific Individual Cognitive Remediation Program in Parkinson's Disease). Group of patients profiting from a structured program of preoperative cognitive remediation
  Interventions: Behavioral: Social adaptation; Procedure: Deep brain stimulation
- ICM group: Intensive Care Management (Other): Group of patients profiting from a preoperative non structured support
  Interventions: Behavioral: Intensive care management; Procedure: Deep brain stimulation
- CG group: Control Group (Other): No supplementary support
  Interventions: Procedure: Deep brain stimulation

INTERVENTIONS:
Behavioral: Social adaptation — Questionnaire to fill-in.
  The structured program of preoperative cognitive remediation is divided in 3 parts: one interview with the patient to do a building of the subjective theories (difficulties due to the disease, hope relative to the intervention), a study meeting of the cognitive remediation possibilities and a cognitive remediation meeting with the patient. The spouse will be included in the program.
  Arms: SICRPPD group
Behavioral: Intensive care management — In this group, the structured program of the SICRPPD group will be replaced by 3 unstructured psychiatric interviews during which patients will be assessed for their perception of the disease and the upcoming surgery. This group will allow to control for the intrinsic effect of the preoperative management independently of the remediation itself.
  Arms: ICM group: Intensive Care Management
Procedure: Deep brain stimulation

SUMMARY:
Main objective:

To assess the impact of a structured program of preoperative cognitive remediation on postoperative social adaptation in patients suffering from Parkinson's disease profiting from bilateral subthalamic nucleus stimulation.

Secondary objectives:

To assess in the same patients the impact of structured program of preoperative cognitive remediation on quality of life, mood, anxiety, apathy and psychologic, social and professional functioning depending on psychiatric symptomatology after intervention.

DETAILED DESCRIPTION:
Prospective, longitudinal, controlled, multicentric, randomised, open study.

Subjects: 3 groups of 40 patients (n=120): one group of patients profiting from a structured program of preoperative cognitive remediation (SICRPPD group: Specific Individual Cognitive Remediation Program in Parkinson's Disease), one group of patients profiting from a preoperative non structured accompaniment (ICM group: Intensive Care Management), one control group (CG group: Control Group).

Required sample size: The sample size of 40 patients/group will allow to demonstrate with a significance threshold of 5% and a power of 80% a difference of evolution of the global SAS SR score of 0.75 SD between 2 of the 3 groups. For an intended SD of 0.2 units, the threshold corresponds to a difference of 0.15 units, minimal significant change.

Intervention: The structured program of preoperative cognitive remediation is divided in 3 parts: one interview with the patient to do a building of the subjective theories (difficulties due to the disease, hope relative to the intervention), a study meeting of the cognitive remediation possibilities and a cognitive remediation meeting with the patient. The spouse will be included in the program.

Evaluation tools: Patients will be met before and after the intervention for clinical evaluations and scales making: For the psychiatric evaluation: Mini International Neuropsychiatric Inventory (M.I.N.I.), Starkstein Apathy Scale, Montgomery and Asberg depression scale (MADRS), global functioning evaluation scale (EGF) and Hamilton anxiety scale (HAMA)/ For the social adaptation evaluation: Social Adjustment scale Self Report (SAS SR)/ For quality of life evaluation: 39-item Parkinson's Disease Questionnaire (PDQ-39)/ For the daily life activities, 'motor' symptomatology and treatment complications evaluation: Unified Parkinson's Disease Rating Scale (UPDRS, parties II, III, et IV).

Main criteria: change in the global score of the SAS SR scale.

Secondary Criteria: change in scores of the PDQ-39 (quality of life), HAMA (anxiety), Starkstein (apathy), MADRS (mood), EGF (psychologic, social, professional functioning, and depending on the psychiatric symptomatology) questionnaires.

Statistics: parametric and non parametric tests will be done for p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Men or women suffering from idiopathic Parkinson's disease for which the indication of treatment by deep cerebral stimulation is retained
* Obtained informed consent

Exclusion Criteria:

* Absence of social security
* Patient unable to be compliant
* Major patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2009-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Global score of the SAS SR (social adjustment scale self report) scale | 3 months (after surgery)
Global score of the SAS SR (social adjustment scale self report) scale | 6 months (after surgery)

SECONDARY OUTCOMES:
Quality of life | 3 months
  evaluated with PDQ-39 (39-item Parkinson's Disease Questionnaire)
Quality of life | 3 months
  evaluated with WHOQOL-bref (World Health Organization Quality of Life)
Quality of life | 6 months
  evaluated with PDQ-39 (39-item Parkinson's Disease Questionnaire)
Quality of life | 6 months
  evaluated with WHOQOL-bref (World Health Organization Quality of Life)
Anxiety | 3 months
  evaluated with HAMA (Hamilton Anxiety Rating Scale)
Anxiety | 6 months
  evaluated with HAMA (Hamilton Anxiety Rating Scale)
Apathy | 3 months
  evaluated with Starkstein scale
Apathy | 6 months
  evaluated with Starkstein scale
Mood | 3 months
  evaluated with Montgomery-Åsberg depression rating scale
Mood | 6 months
  evaluated with Montgomery-Åsberg depression rating scale
Global Assessment of Functioning | 3 months
  to rate the social, occupational, and psychological functioning according to psychiatric symptomatology
Global Assessment of Functioning | 6 months
  to rate the social, occupational, and psychological functioning according to psychiatric symptomatology
Disease perception | 3 months
  Illness Perception Questionnaire Revised
Disease perception | 6 months
  Illness Perception Questionnaire Revised
Perception of deep brain stimulation | 3 months
  with Perception of deep brain stimulation scale
Perception of deep brain stimulation | 6 months
  with Perception of deep brain stimulation scale
Coping with disease | 3 months
  with CHIP scale
Coping with disease | 3 months
  with Brief COPE scale
Coping with disease | 6 months
  with CHIP scale
Coping with disease | 6 months
  with Brief COPE scale

CONTACTS AND LOCATIONS:
Overall Officials: Raymund Schwan, Prof., Principal Investigator — Nancy's Hospital; Gérard Barroche, Prof., Principal Investigator — CHU of Nancy - Central Hospital - Bd Marechal de Lattre de Tassigny - 54000 Nancy; Marie-Christine Tranchant, Prof., Principal Investigator — CHU of Strasbourg - 67000 Strasbourg; Franck Durif, Prof, Principal Investigator — CHU Clermont-Ferrand - 63000 Clermont Ferrand
Locations (3):
- France (3):
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU de Nancy, Nancy
  - CHRU Strasbourg, Strasbourg

REFERENCES:
- [Derived] Meyer M, Colnat-Coulbois S, Frismand S, Vidailhet P, Llorca PM, Schwan R, Spitz E. Illness perceptions in pre-operative Parkinson's disease patients. J Neural Transm (Vienna). 2023 May;130(5):647-654. doi: 10.1007/s00702-023-02629-2. Epub 2023 Apr 6. PMID 37022502